CLINICAL TRIAL: NCT00690807
Title: A Phase 2 Efficacy and Safety Study of PH-10 Aqueous Hydrogel for the Treatment of Atopic Dermatitis
Brief Title: A Phase 2 Study of PH-10 for the Treatment of Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Provectus Pharmaceuticals (Industry)
Responsible Party: Eric Wachter, Vice President, Provectus Pharmaceuticals, Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH-10-AD-21
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2009-09-28 (Estimated); Status verified 2009-09

CONDITIONS: Atopic Dermatitis
Keywords: eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): PH-10 treatment
  Interventions: Drug: PH-10

INTERVENTIONS:
Drug: PH-10 — PH-10 will be applied daily for 28 days to skin areas affected by atopic dermatitis.

SUMMARY:
PH-10 is a formulation of rose bengal disodium (RB) for topical administration to the skin. PH-10 is capable of undergoing photochemical reactions when activated by ambient light. This phase 2 study will assess whether topical PH-10 applied once daily to mild, moderate or severe areas of atopic dermatitis (including atopic eczema) may ameliorate inflammation of the skin when activated by ambient light.

ELIGIBILITY:
Inclusion Criteria:

* Men or women, age 18 or older.
* Mild, moderate or severe atopic dermatitis.
* Presence of atopic dermatitis areas outside the head and face with a baseline Investigator Global Assessment (IGA) of 2 (mild disease), 3 (moderate) or 4 (severe disease) at screening.
* Written informed consent by the subject or legal guardian.

Exclusion Criteria:

* Women who are pregnant, attempting to conceive, or nursing an infant.
* Subjects who have received phototherapy (UVB, PUVA) or systemic therapy (immunosuppressants, cytostatics, corticosteroids) within 4 weeks.
* Subjects who have received systemic antibiotics within 2 weeks.
* Subjects who have received topical therapy (tar, corticosteroids) within 7 days.
* Subjects who have received investigational drugs in a clinical research study within 4 weeks.
* Subjects who have received agents posing a clinically significant risk of photosensitivity reaction within 5 half-lives of initiation of study treatment.
* Subjects with a history of porphyria, systemic lupus erythematosus or xeroderma pigmentosum.
* Subjects with clinical conditions that may pose a health risk to the subject by being involved in the study or detrimentally affect regular follow-up of the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-06; Primary Completion 2009-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is "Treatment Success," a static endpoint defined as a score of 0 to 1 at Day 28 (at the end of the study treatment period) by the Investigator's Global Assessment (IGA) scoring system for atopic dermatitis status. | 28 days
Adverse experience, including pain and dermatologic/skin toxicity (incidence, severity, frequency, duration and causality). | 8 weeks

SECONDARY OUTCOMES:
Investigator's Global Assessment (IGA) score changes at each visit from Day 1 pre-treatment. | 8 weeks
Eczema Area Severity Index (EASI) score changes of individual atopic dermatitis signs at each visit from Day 1 pre-treatment. | 8 weeks
Pruritus Self-Assessment score changes of atopic dermatitis related itching/scratching at each visit from Day 1 pre-treatment. | 8 weeks
Adverse change in clinical laboratory tests (CBC and CMP). | 8 weeks
Adverse change in vital signs (BP, pulse, temperature). | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alicia Barba, MD, Principal Investigator — International Dermatology Research, Inc.
Locations (2):
- United States (2):
  - International Dermatology Research, Miami, Florida
  - Mount Sinai School of Medicine, New York, New York